CLINICAL TRIAL: NCT03018314
Title: Serum Kisspeptin Levels in Infertile Women Due to Anovulatory Cycles, Unexplained Infertility or Male Subfertility: A Prospective Observational Study
Brief Title: Serum Kisspeptin Levels in Infertile Women
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016/165
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Infertility, Female; Unexplained Infertility; Anovulation
MeSH Terms: conditions — Infertility, Female; Anovulation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: The first group will comprise of 30 women with polycystic ovaries in ultrasound examination or anovulatory cycles.
  Interventions: Other: Blood sample
- Group 2: The second group will comprise of 30 women with diagnosis of unexplained infertility, normal menstrual periods and without known male factor infertility.
  Interventions: Other: Blood sample
- Group 3: The third group will comprise of 30 women those partners with sperm count between 5x106 -15x106 /mL, type A + type B motility <%32 and Kruger morphology <4%.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Serum analysis
  Other Names: Serum Kisspeptin levels

SUMMARY:
The study population is comprise of 90 women those age varies between 18-38 year-old. The first group will comprise of 30 women with polycystic ovaries or anovulatory cycles, the second group will comprise of 30 women with diagnosis of unexplained infertility and the third group will comprise of 30 women those partners with male subfertility. A 2 cc blood sample for Kisspeptin analysis will be drawn from the antecubital vein from each participants. The patients will receive 50 mg clomiphene citrate at the fifth day of the menstrual period and follicular development will be measured with serial ultrasound follow up.

DETAILED DESCRIPTION:
The study population is comprise of 90 women those age varies between 18-38 year-old with wish of baby for at least one year despite of unprotected sexual intercourse, patent tubes confirmed in hysterosalpingography , follicle stimulating hormone levels <12 IU. The first group will comprise of 30 women with polycystic ovaries in ultrasound examination or anovulatory cycles, the second group will comprise of 30 women with diagnosis of unexplained infertility, normal menstrual periods and without known male factor infertility and the third group will comprise of 30 women those partners with sperm count between 5x106 -15x106 /mL, type A + type B motility <%32 and Kruger morphology <4%. A 2 cc blood sample for Kisspeptin analysis will be drawn from the antecubital vein from each participants and centrifuged and sera will be kept in -80 C till recruitment has been completed. Kisspeptin, E2, Progesterone, anti-mullerian hormone levels will be measured with ELISA method. The patients will receive 50 mg clomiphene citrate at the fifth day of the menstrual period and follicular development will be measured with serial ultrasound follow up.

ELIGIBILITY:
Inclusion Criteria:

* ages varying between 18-38 year-old with wish of baby for at least one year despite of unprotected sexual intercourse
* patent tubes confirmed in hysterosalpingography
* follicle stimulating hormone levels <12 IU
* no other relevant medical history

Exclusion Criteria:

* ages other than 18-38 year-old with wish of baby for least than one year despite of unprotected sexual intercourse
* obstructed tubes confirmed in hysterosalpingography
* follicle stimulating hormone levels >12 IU
* history thyroid disease
* increased prolactin levels
* history of chemo/radiation therapy

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 90 infertile female women those with infertile couples due to anovulation,male sub fertility and unexplained infertility.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The relation of Kisspeptin levels and female infertility | 1 year

SECONDARY OUTCOMES:
The relation of Kisspeptin levels and follicular growth | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Kaya, M.D., Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After study completed

REFERENCES:
- [Background] Skorupskaite K, George JT, Anderson RA. The kisspeptin-GnRH pathway in human reproductive health and disease. Hum Reprod Update. 2014 Jul-Aug;20(4):485-500. doi: 10.1093/humupd/dmu009. Epub 2014 Mar 9. PMID 24615662
- [Derived] Kaya C, Alay I, Babayeva G, Gedikbasi A, Ertas Kaya S, Ekin M, Yasar L. Serum Kisspeptin levels in unexplained infertility, polycystic ovary syndrome, and male factor infertility. Gynecol Endocrinol. 2019 Mar;35(3):228-232. doi: 10.1080/09513590.2018.1519792. Epub 2018 Oct 17. PMID 30328739
- See also: PUBMED — https://www.ncbi.nlm.nih.gov/pubmed/?term=The+kisspeptin-GnRH+pathway+in+human+reproductive+health+and+disease